CLINICAL TRIAL: NCT04793360
Title: Molecular Assessment and Profiling of Liver Transplant Recipients
Acronym: MAPLE
Status: Active, not recruiting | Type: Observational
Sponsor: CareDx (Industry)
Responsible Party: Sponsor
Other Study IDs: SN-C-00015
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Liver Transplantation; Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LiverCare Surveillance: Participants undergoing orthotopic liver transplant (de-novo or re-transplant) will be considered for this study
  Interventions: Device: LiverCare

INTERVENTIONS:
Device: LiverCare — The LiverCare kits contains Streck tubes and PAX gene tubes, which will be collected at the surveillance schedule outlined above, but also prior to any liver biopsy or DSA measurement. For patients who have a histological diagnosis of allograft rejection who are undergoing treatment, serial monitoring of LiverCare will be performed following the schedule above. All research blood tests will be timed with standard clinical testing to avoid any additional needle sticks.

SUMMARY:
The objective of this protocol is to conduct longitudinal and prospective studies of liver transplant recipients, using a multimodality approach, akin to that used in kidney transplantation. The primary aim will compare the clinical outcomes of LiverCare post-transplant surveillance in liver transplant with standard of care consisting of liver function tests, DSA measurements, drug level monitoring, and 'for cause' biopsy. The protocol will assess the correlation between clinical events (e.g. rejection, recurrent disease, biliary obstruction), dd-cfDNA levels, gene expression profiling, ability to assess microchimerism, develop predictive analytics, infectious disease diagnoses and finally examine graft histology.

ELIGIBILITY:
Inclusion Criteria:

* Liver transplant recipients <60 days post-transplant (de-novo or re-transplant).
* Participant is willing and able to give informed consent for participation in the trial.
* Male or Female, aged 12 years or above (Gillick Competent).
* In the Investigator's opinion, is able and willing to comply with all trial requirements.

Exclusion Criteria:

* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial.
* Has evidence of significant post-transplant impairment of hepatic function which is unlikely to improve (determined by the PI).
* Scheduled elective surgery or other procedures requiring general anaesthesia during the trial.
* Participant with life expectancy of less than 6 months or is inappropriate for diagnostic monitoring through regular blood sampling.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Participants who have participated in another research trial involving an investigational product in the past 12 weeks*.
* Multi-organ transplant recipients or dual organ transplant recipients.
* Patients with significant needle phobia.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All liver transplant patients without exclusion criteria will be eligible to enter the study. Patients will be approached by the study team at the time of transplant or within 60 days post-transplant to discuss the trial, consent and enrollment.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
To correlate the results of LiverCare with clinically significant events impacting post-transplant clinical outcomes, histological findings, and the development of de novo Donor Specific Antibody (DSA) | 2 years of accrual and 3 years follow up
  LiverCare will be measured 7 times in year 1 and quarterly each year. A total of 15 surveillance points per subject in addition to for-cause testing based on clinical changes. Liver care will be collected at the time of all histologic analyses whether 'for cause' or 'surveillance'

CONTACTS AND LOCATIONS:
Overall Officials: Kanish Mohib, PhD, Study Director — CareDx
Locations (26):
- United States (26):
  - Keck Medical Center of USC, Los Angeles, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Tampa General Hospital, Tampa, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - Tulane University, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (BIDMC), Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Washington Unversity in St. Louis, St Louis, Missouri
  - University of Nebraska Medical Center/ Nebraska Medicine, Omaha, Nebraska
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Westchester Medical Center, Valhalla, New York
  - Atrium Health, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - INTEGRIS Baptist Medical Center, Oklahoma City, Oklahoma
  - Medical Unversity of South Carolina, Charleston, South Carolina
  - University of Tennessee_Methodist Healthcare, Memphis, Tennessee
  - Methodist Health System, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle, Washington